CLINICAL TRIAL: NCT00178308
Title: Measuring Alterations of DNA in Human Blood
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Litron Laboratories (Industry)
Other Study IDs: URCC 1702
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purpose of this research is to evaluate an automated, laser-based technique for measuring DNA damge resulting from radiation. We want to use controlled exposure on cancer patients to help develop a measurement to test people who may have been accidentally exposed to radiation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 21 to 70 years old.
* Patient undergoing with anti-neoplastic agent(s) known to have genotoxic activity (e.g., cyclophosphamide, 5-FU, cisplatin, Ara-C.
* X-irradiation may be considered, so long as a substantial fraction of red marrow is exposed (e.g., femur or chest/trunk region);
* treatment could be ongoing therapy or initial therapy.

Ages: 21 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 24

CONTACTS AND LOCATIONS:
Overall Officials: Yuhchyau Chen, MD, Ph.D, Principal Investigator — Universtiy of Rochester, Dept of Radiation Oncology
Locations (1):
- University of Rochester, Rochester, New York, United States